CLINICAL TRIAL: NCT04630418
Title: NanoSilk Cosmo: Evaluation of a Novel Silk Complex on Biophysical Parameters Related to Skin Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-2033
Record Dates: First submitted 2020-10-22; First posted 2020-11-16 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NanoSilk Cosmo (Experimental): Participants will receive a 30 mL jar of NanoSilk Cosmo
  Interventions: Other: NanoSilk Cosmo

INTERVENTIONS:
Other: NanoSilk Cosmo — Participant will receive 30 mL of NanoSilk Cosmo jar.

SUMMARY:
Silk is a naturally occurring protein polymer that is approved for medical use by the U.S Food and Drug Administration (FDA). Silk fibroin fiber biomaterial has shown promising results for tissue regeneration demonstrated through in vivo and in vitro animal models. The investigators of this study have previously shown that patients' report improvement in common skin aging findings including wrinkles, sagginess, and dry skin. The investigators will continue this assessment of patients' skin perception as well as add on objective measures of skin resilience, elasticity, and hydration.

The investigators will provide participants with a demographic survey, and the FACE-Q survey, a validated survey, prior to administration of NanoSilk Cosmo, to assess perception of aging, satisfaction with facial appearance, satisfaction with skin. The participant will undergo baseline evaluation of several objective measures of skin hydration, elasticity and overall healthy using non-invasive devices (Courage+Khazaka Corneometer Probe, Courage+Khazaka Electronic GmbH Cutometer Dual MPA 580, and VISIA-CA GEN 7). The participants will be provided with 30ml of the NanoSilk Cosmo and with extensive instruction on administration of the product.

Participants will return to clinic after 4 weeks of using the product to perform the FACE-Q and re-evaluation of several objective measures of the skin using non-invasive devices (Courage+Khazaka Corneometer Probe, Courage+Khazaka Electronic GmbH Cutometer Dual MPA 580, and VISIA-CA GEN 7).

DETAILED DESCRIPTION:
Skin aging is characterized by atrophy, decreased elasticity, wrinkling, impaired strength, and altered metabolic and reparative responses. The etiology of these changes is multifactorial and includes intrinsic factors such as age, genetics, metabolism, and nutrition, as well as extrinsic or environmental effects like Ultraviolet (UV) radiation and air pollution. It has been noted that there is increased fragility of the skin with age due to flattening of the dermo-epidermal junction and decreased biosynthetic capacity of fibroblasts, all leading to decreased skin resilience and an undesirable cosmetic appearance of the skin.

Recently, the use of silk to reverse or repair some of these aging processes has gained significant interest. Silk is a natural protein polymer that is approved for medical use by the U.S. Food and Drug Administration and Bombyx mori (B. mori) silk is considered a non-animal product (EU Council Directive 93/42/EEC, rule 17). Importantly it is biocompatible, non-inflammatory, and non-cytotoxic. There are two important components of silk that are derived from the B. mori worm, both of which are proteins - fibroin and sericin. In simple terms, sericin, which represents about 30% of the entire cocoon, functions as a glue to hold the fibroin fibers together while blocking UV rays and providing moisture. The fibroin, approximately 70% of the cocoon, is composed of two proteins which interestingly have similar amino acid compositions to Natural Moisturizing Factor which is found in the stratum corneum of human skin and helps retain moisture in the skin. The stratum corneum is of key importance to the skin's ability to hold water and maintain skin integrity which is critical for maintaining a youthful appearance.

Besides the moisture retention effects noted above, one of the theories behind the effectiveness of silk on the skin is that the silk fibroin nanofibers are able to promote cell adhesion and allows type I collagen to spread within epidermal keratinocytes and fibroblasts. New data suggest that if a patient has a higher ratio of collagen type I to collagen type III that these patients will have better outcomes after aesthetic facial surgery, which highlights the key role of collagen in the skin.

The investigators will provide participants with the FACE-Q survey, a validated survey, prior to administration of NanoSilk Cosmo, to assess perception of aging, satisfaction with facial appearance, and satisfaction with skin. The participant will undergo baseline evaluation of several objective measures of skin hydration, elasticity and overall healthy using non-invasive devices (Courage+Khazaka Corneometer Probe, Courage+Khazaka Electronic GmbH Cutometer Dual MPA 580, and VISIA-CA GEN 7). The participants will be provided with 30ml of the NanoSilk Cosmo and with extensive instruction on administration of the product.

Participants will return to clinic after 4 weeks of using the product to perform the FACE-Q and re-evaluation of several objective measures of the skin using non-invasive devices (Courage+Khazaka Corneometer Probe, Courage+Khazaka Electronic GmbH Cutometer Dual MPA 580, and VISIA-CA GEN 7).

Courage+Khazaka Corneometer Probe: By evaluating the capacitance through the skin this will serve as a reflection of moisture content in the skin. The corneometer is not significantly affected by stales or residues of topicals applied to the skin. Additionally, it provides very quick measurements (1 sec), continuous measurements, and the measurement depth is very small to capture the stratum corneum and avoid deeper skin structures (blood vessels). The Visioscan measures an integral characteristic of skin, and included metric in the clinical experiment. It is medical grade (degree of calibration) and will provide the most accurate data for researchers.

The probe will be placed on the skin before and after use of NanoSilk Cosmo and measure the data points noted above.

Courage+Khazaka Electronic GmbH Cutometer dual MPA 580: This device will measure viscoelasticity of the skin using negative pressure to mechanically deform the skin. The penetration depth is determined by a non-contact optical measuring system within the probe. The resistance of the skin to the negative pressure (firmness) and its ability to return to its original position (elasticity) are displayed as curves (penetration depth in mm/time) in real time. The measurement allows for information about the elastic and mechanical properties of skin surface and to objectively quantify a property of skin aging. The Cutometer measures an integral characteristic of skin and included metric in the clinical experiment. It is medical grade (degree of calibration) and will provide the most accurate data for researchers.

The probe will be placed on the skin before and after use of NanoSilk Cosmo and measure the data points noted above.

VISIA-CA GEN 7(Consultation System): VISIA multi-point positioning system and live image overlay provides complete data surface and subsurface skin conditions. Skin conditions included in analysis are hyperpigmentation, hypopigmentation, inflammation, wrinkles, topography, UV damage, vascularity (spider veins), and porphyrins.

The participant will place their face in the instrument and have their photo taken both before and after use of NanoSilk Cosmo.

ELIGIBILITY:
Inclusion Criteria:

* Male, female, and gender non-binary
* Age 18 years and older
* Any race or ethnicity
* Those with evidence of age-related skin changes.

Exclusion Criteria:

* <18 years of age
* Pregnant
* Decisionally challenged

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Subjective patient perception of skin | 6 months
  Evaluate patient's perception of satisfaction with skin before and after application of NanoSilk Cosmo using surveys designed to target and answer these questions. Copies of these surveys are below.
  Scale Titles: NanoSilk Cosmo Initial Survey and NanoSilk Cosmo Completion Survey
  There are no minimum or maximum values of this scale, therefore there is no high or low score. This is a scale to determine the demographics and use patterns of those who use NanoSilk Cosmo. Additionally, it will give the option for feedback on the product and ask participants to evaluate the effect the product had on their skin.
Change in skin hydration levels | 6 months
  To perform a prospective clinical trial to quantitatively assess the effects of NanoSilk Cosmo solution on the hydration status of the skin using the Courage + Khazaka Electronic Corneometer which uses a capacitance measurement of a dielectric medium that changes with increased or decreased hydration in the stratum corneum layer of the skin.
Change in skin viscoelasticity levels | 6 months
  To perform a prospective clinical trial to quantitatively assess the effects of NanoSilk Cosmo solution on the viscoelasticity of the skin using the Courage + Khazaka Electronic GmbH Cutometer which uses negative pressure to deform the skin and then measures its ability to return to the original position. These measurements are then displayed on a curve for which normal skin has been previously established.
Change in skin surface topography | 6 months
  To perform a prospective clinical trial to quantitatively assess the effects of NanoSilk Cosmo solution on the skin surface topography using VISIA Gen 7. This device uses a non-invasive photograph and then through a series or different lighting on this photograph evaluates common skin surface topography concerns such as spots, pores, wrinkles, texture, porphyrins, UV spots, red areas, and brown spots.

CONTACTS AND LOCATIONS:
Overall Officials: Brooke French, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Health and Wellness Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No